CLINICAL TRIAL: NCT05337332
Title: Suprachoroidal Triamcinolone Acetonide Injection in Two Chorioretinal Diseases: One Year Results
Brief Title: Results of Suprachoroidal Steroids Injections in Two Chorioretinal Diseases
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Assistant professor of Ophthalmology, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 7-7-22
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Central Serous Chorioretinopathy; Irvine-Gass Syndrome; Pars Planitis; Cystoid Macular Edema
Keywords: Central serous chorioretinopathy; Cystoid macular edema
MeSH Terms: conditions — Central Serous Chorioretinopathy; Macular Edema; Pars Planitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Central serous chorioretinopathy group (Experimental): Cases with central serous chorioretinopathy (CSR) that will be injected with suprachoroidal triamcinolone acetonide.
  Interventions: Drug: Triamcinolone Acetonide
- Irvine-Gass Syndrome group (Experimental): Cases with cystoid macular edema due to irvine-gass syndrome that will be injected with suprachoroidal triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Suprachoroidal injection of triamcinolone acetonide
  Other Names: Suprachoroidal triamcinolone acetonide injection (SCTA)

SUMMARY:
Suprachoroidal injection is a safe way for intraocular drug delivery. It was used to treat various retinal conditions.

DETAILED DESCRIPTION:
Suprachoroidal triamcinolone acetonide injection is used to treat various retinal diseases, higher concentration of the injected material is found when the suprachoroidal space is used as an intraocular delivery pathway when compared to the conventional intravitreal pathway.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed as central serous chorioretinopathy and patients with cystoid macular edema due to irvine-gass syndrome after cataract surgery.

Exclusion Criteria:

* other retinal diseases that may affect CMT and final visual outcome.
* Patients with dense corneal opacity.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Central macular thickness | Baseline and 12 months after injection.
  Changes in central macular thickness (CMT) measured in millimeters (mm) by optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Best corrected visual acuity | Baseline and 12 months after injection.
  Changes in best corrected visual acuity (BCVA) measured in logarithm of minimal angle of resolution (LogMAR) by chart projector.

OTHER OUTCOMES:
Intraocular pressure | Baseline and 12 months after injection.
  Changes in intraocular pressure (IOP) measured in millimeter mercury (mmHg) by applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelshafy, MD, Principal Investigator — Benha University
Locations (1):
- Ahmed Abdelshafy, Banhā, QA, Egypt

IPD SHARING:
Plan to Share IPD: No